CLINICAL TRIAL: NCT00517088
Title: Level of Physical Activities in Patients Before and After Breast Cancer Treatment
Acronym: PABC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UPECLIN HC FM Botucatu Unesp (Other)
Allocation: Not Applicable | Model: Single Group | Masking: Single
Other Study IDs: upeclin/HC/FMB-Unesp-pre03
Expanded Access: Available
Record Dates: First submitted 2007-08-14; First posted 2007-08-16 (Estimated); Last update posted 2014-05-30 (Estimated); Status verified 2007-08

CONDITIONS: Breast Cancer
Keywords: Physical Activity; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Other (Other): Group Description
  Interventions: Drug: IPAQ

INTERVENTIONS:
Drug: IPAQ

SUMMARY:
Subjects and Methods: 303 patients who had already had the diagnosis of breast cancer and had already been treated at the Ambulatory of Botucatu School of Medicine were selected. The measuring tool used for the level of physical activities was the International Physical Activities Questionnaire (IPAQ-short version), validated by the World Health Organization - Physical Activities and Health International Committee (1998).

DETAILED DESCRIPTION:
Introduction: Breast cancer is the most common malignant neoplasy in women. The risk for breast cancer in a lifetime is high among north-american women, about one out of eight, with 66% of the cases occurring after menopause and 15% when women are under 40 years old. Published cohort studies show clear evidences that women who practice intense physical activities have the risk for breast cancer reduced. The risk reduction for these women is 70%, and 10% for those who practice physical activities at a low level. During adolescence and adult age, moderate to intense physical activities may protect against a future breast cancer development. But some questions still need to be answered: Were women with a breast carcinoma diagnosis already physically active during life? Were there changes in these physical activities after treatment? Why? Objectives: The aim of this study was to identify the level of physical activities in patients before and after breast carcinoma treatment, and to observe if there were changes in the level of these activities. Subjects and Methods: 303 patients who had already had the diagnosis of breast cancer and had already been treated at the Ambulatory of Botucatu School of Medicine were selected. The measuring tool used for the level of physical activities was the International Physical Activities Questionnaire (IPAQ-short version), validated by the World Health Organization - Physical Activities and Health International Committee (1998).

ELIGIBILITY:
Inclusion Criteria:

* Patients whit diagnosis of breast cancer

Ages: 20 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2007 (Actual)
Dates: Start 2006-05; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
breast cancer | one year

CONTACTS AND LOCATIONS:
Overall Officials: Flávio G Pinto, Principal Investigator — UPECLIN HC FM Botucatu Unesp